CLINICAL TRIAL: NCT04785872
Title: EFFECT OF NEUMAN SYSTEMS MODEL BASED NURSING APPROACH ON STRESS AND COPING WITH STRESS FOR WOMEN RECEIVED INTRAUTERIN INSEMINATION TREATMENT
Brief Title: Neuman Systems Model and Infertility Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Menekşe Nazlı AKER, Lecturer, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16726501
Record Dates: First submitted 2021-02-28; First posted 2021-03-08 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Infertility; Intrauterine Insemination
MeSH Terms: conditions — Infertility | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: Education
- Control group (No Intervention)

INTERVENTIONS:
Other: Education — NEUMAN SYSTEMS MODEL BASED NURSING APPROACH
  Other Names: Relaxation
  Arms: Intervention group

SUMMARY:
In this study, it is aimed to determine the effect of Neuman Systems Model based nursing approach on stress an coping with stress for women received intrauterine insemination (IUI) treatment. The study has been planned as a single blind experimental study in pretest-posttest design with randomized control. Sample group is going to be chosen from women who have taken IUI treatment in Ankara University Fertility Diagnosis, Treatment, Research and Application Center. Sample size of the study has been determined as 72 such that intervention=36 and control=36. While gathering data, personal information form, The COMPI Fertility Problem Stress Scales and The COMPI Coping Strategy Scales are going to be used. In the scope of the study, four interviews with women in intervention group are going to be done during IUI treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Getting a diagnosis of primary infertility
2. Volunteering to participate in the study
3. Being over the age of 18
4. Taking IUI treatment
5. Not being diagnosed with a chronic disease
6. Not being diagnosed with a psychiatric illness
7. Do not have a problem that can interfere with written and verbal communication.

Exclusion Criteria:

1. To want to leave the study,
2. Cancellation of treatment.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2020-10-19 (Actual); Study Completion 2020-10-19 (Actual)

PRIMARY OUTCOMES:
The COMPI Fertility Problem Stress Scale | Immediately after intrauterine insemination procedure
  The scale is used for the assessment of the levels of stress experienced by infertile couples. As a Likert-type scale, it has three sub-scales in relation to personal, marital and social domains and contains a total of 14 items. 'Stress in personal domain' sub-scale contains six items, and the minimum and maximum scores to be obtained from it are successively 0 and 20 points. 'Stress in marital domain' sub-scale has four items, and the minimum and maximum scores to be obtained from it are successively 0 and 14 points. 'Stress in social domain' sub-scale is comprised of four items, and the minimum and maximum scores to be obtained from it are successively 0 and 12 points. A high score to be obtained from the sub-scale refers to the increase in the stress level.
The COMPI Coping Strategy Scale | Immediately after intrauterine insemination procedure
  The scale contains 19 items and has four sub-scales. The minimum and maximum scores to be obtained from the sub-scale of 'active-avoidance' coping method which is comprised of four items are successively 4 and 16 points. The sub-scale of 'active-confronting' coping method contains seven items. The minimum and maximum scores to be obtained from this sub-scale are successively 7 and 26 points. The minimum and maximum scores to be obtained from the sub-scale of 'passive-avoidance' coping method which is comprised of three items are successively 3 and 12 points. The sub-scale of 'meaning-based' coping method contains five items. The minimum and maximum scores to be obtained from this sub-scale are successively 5 and 20 points. A higher score to be obtained from the subscale means that the method is used more when coping with with stress.

CONTACTS AND LOCATIONS:
Overall Officials: Menekşe N Aker, PhD, Study Chair — Ankara University Nursing Faculty
Locations (1):
- Ankara University Fertility Diagnosis, Treatment, Research and Application Center, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No